CLINICAL TRIAL: NCT06866392
Title: Study on Novel Strategies for Cervical Cancer Screening Using Photoelectric Detection Combined with Epigenetic Procotol
Brief Title: Study on Novel Strategies for Cervical Cancer Screening Using Photoelectric Detection and Epigenetic Procotol
Acronym: CC-AZ
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CCAZ
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group: Methylation test and colposcopic biopsy, and clinical follow-up based on methylation results
- OITS group: The experimental group underwent methylation test and colposcopic biopsy and OITS, and clinical follow-up was conducted according to methylation results and OITS results
  Interventions: Diagnostic Test: photoelectric detection

INTERVENTIONS:
Diagnostic Test: photoelectric detection — Methylation test and colposcopic biopsy was performed in the conventional group, and clinical follow-up was performed according to the methylation results; in the experimental group, methylation test and colposcopic biopsy and OITS was performed, and clinical follow-up was performed according to the methylation results and OITS results.
  Groups: OITS group

SUMMARY:
A national multicenter, open randomized controlled study was conducted. It is planned to invite 30 multi-center units across the country to compete for enrollment, and each multi-center will enroll 140 patients meeting colposcopic indications (70 in the conventional group and 70 in the experimental group), totaling 4200 patients. Enrolled subjects were randomly divided into two groups. Methylation test + colposcopic biopsy was performed in the conventional group, and clinical follow-up was performed according to the methylation results; in the experimental group, methylation test + colposcopic biopsy +OITS was performed, and clinical follow-up was performed according to the methylation results and OITS results. To verify the effectiveness of methylation tests and OITS in screening for CIN2+, whether they can reduce missed diagnosis of CIN2+, whether they can flag excessive colposcopic procedures, and the value of clinical follow-up for cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 18 and 65 who have already had sex life
2. HPV16, 18 positive or high-risk HPV infection with cytology ≧ASC-US
3. No history of cervical cancer and cervical physical therapy, a complete cervix
4. No menstrual period, no sexual activity and vaginal medication within 48 hours
5. The vagina or cervix is not in a stage of acute inflammation
6. Willing to participate in the study with full informed consent

Exclusion Criteria:

1. Cervical dysplasia (congenital malformation or double uterus, etc.)
2. History of cervical treatment (coning, ablation, or photodynamic therapy)
3. There are definite immunosuppression conditions, such as HIV infection or organ transplantation
4. Patients with severe bleeding diseases such as coagulation abnormalities or photosensitive diseases (such as porphyria, lupus erythematosus, etc.)
5. A history of radiation or chemotherapy (e.g., pelvic radiation therapy) with cancer at other sites
6. The patient is in pregnancy or puerperium
7. The other conditions of this study were not considered appropriate by the researchers

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 30 multi-center units in the country, and each center competes to enter the group. The accuracy of OITS early data was 75%, the sensitivity was 82%, and the specificity was 63%. According to 20% shedding, possible causes of shedding: error caused by severe inflammatory patients, error caused by improper operation or subjects unwilling to cooperate with follow-up. The optimal efficacy test was performed with the rate of 0.75 in the experimental group and 0.5 in the control group, and the optimal efficacy threshold was 0.1(control-experimental group), bilateral alpha was 0.05, beta was 0.2, and the sample size ratio of the two groups was 1(experimental group: Control group), each single center needs to collect 58 cases in the experimental group and 58 cases in the control group. Considering 20% shedding, the sample size of each single center is at least 70 cases in the experimental group and 70 cases in the control group, and a total of 4200 cases of all centers.
Sampling Method: Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of a photoelectric image detector for cervical lesions | Enrolled subjects receive histopathological results approximately 7 days after colposcopy
  Sensitivity and specificity of the photoelectric detection technique relative to histopathological findings.

SECONDARY OUTCOMES:
Detection rate of CIN2+ by photoelectric cervical lesion image detector | Enrolled subjects receive histopathological results approximately 7 days after colposcopy.
  The sensitivity, specificity, CIN2+ detection rate, negative predictive value and positive predictive value were compared with the results of Methylaiton, colpscopy, HPV detection and cytology.